CLINICAL TRIAL: NCT04728685
Title: Effects of One-fifth, One-third, and One-half of the Bodyweight Lumbar Traction on the Straight Leg Raise Test and Pain in Prolapsed Intervertebral Disc Patients
Brief Title: Effects of Lumbar Traction on the Straight Leg Raise Test and Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRC-2019-29
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Prolapsed Intervertebral Disc
Keywords: Mechanical Traction; Prolapsed intervertebral disc; straight leg raise test; pain
MeSH Terms: conditions — Intervertebral Disc Displacement; Pain

STUDY DESIGN:
Intervention Model Description: Three-arm parallel groups
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): One-fifth of body weight traction force will be given
  Interventions: Procedure: Mechanical Traction
- Group B (Active Comparator): One-third of body weight traction force will be given
  Interventions: Procedure: Mechanical Traction
- Group C (Active Comparator): One-half of body weight traction force will be given
  Interventions: Procedure: Mechanical Traction

INTERVENTIONS:
Procedure: Mechanical Traction — Mechanical Traction will be applied to the lumbar region using a traction unit.

SUMMARY:
Disc prolapse causes impairment of function by nerve root compression compelling the patient to seek medical advice for low backache. Traction is one of the physical modalities frequently used for the treatment of lumbar disc herniations. So the purpose of the study is to determine the effect of one-fifth, one-half, and one-third of body weight traction on the straight leg raise test and pain.

DETAILED DESCRIPTION:
A total of 45 patients suffering from lumbar PIVD and having neurological symptoms will be selected for the study. Lumbar PIVD will be confirmed from MRI. Participants will be divided into three groups with 15 participants in each group. group A. for one-fifth of body weight traction, group b for one-third of body weight traction, and group C for one-half of body weight traction. SLR and pain will be measured before traction and after traction. A goniometer will be used to measure SLR and VAS will be used to measure pain.

ELIGIBILITY:
Inclusion Criteria:

* Back pain for less than 3 months
* Positive unilateral Straight Leg Raise test which includes reports of back and leg pain or paraesthesia below 45-degree hip flexion
* At least one additional neurological sign should be present including- (a) Diminished Achillis/Hamstring tendon reflex, tested in the supine position or (b) Hyposthesia in any of the L4-S2 dermatome, or (c) Muscle weakness in any of the L4-S2 myotome.
* MRI evidence of L-4-L5 or L5-S1 disc prolapse or both.

Exclusion Criteria:

* Malignancy, Tuberculosis, Osteoporosis, Osteomyelitis of the vertebral column
* Cord compression, Pregnancy, Hypertension, Cardiovascular disease, Joint hyper mobility
* Subjects who could not tolerate the traction force secondary to being in an acute stage of back pain.
* Subjects who have taken previous physiotherapy treatment in the last three months for back pain.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-03-24 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Straight Leg Raise test | upto 1 month
  Straight leg raise test is used in supine position to test neurological signs
Visual analog scale | upto 1 month
  Visual analog scale is used to measure pain. This scale has 0 to 10 points, 0 being no pain and 10 means maximum pain someone has felt. Higher the score worse is the condition.

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, MPTh, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No